CLINICAL TRIAL: NCT07185347
Title: A Randomized, Parallel-arm, Double Blind, Placebo-controlled Study to Assess the Efficacy of Fampridine for Patients With Spinocerebellar Ataxia SCA27B Caused by a GAA Expansion in the FGF14 Gene
Acronym: TREAT-FGF14
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP240921; 2024-520413-53-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-03; First posted 2025-09-22 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Spinocerebellar Ataxia 27B (SCA27B)
Keywords: SCA27B; Fampridine; Ataxia; Diplopia; FARS-Functional Staging
MeSH Terms: conditions — Ataxia; Diplopia | interventions — 4-Aminopyridine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fampridine (Experimental)
  Interventions: Drug: Fampridine 10 mg prolonged-release tablet (per os)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo (tablets per os)

INTERVENTIONS:
Drug: Fampridine 10 mg prolonged-release tablet (per os) — Patients randomized in the experimental arm will take 1 tablet twice a day, 12 hours apart, on an empty stomach, for 12 weeks.
  Arms: Fampridine
Drug: Placebo (tablets per os) — Patients randomized in the control arm will take 1 tablet twice a day, 12 hours apart, on an empty stomach, for 12 weeks.
  Arms: Placebo

SUMMARY:
Spinocerebellar ataxias 27B (SCA27B) is caused by an expansion of ≥ 250 GAA triplets in the FGF14 gene and accounts for 15% of cerebellar ataxias (around 500 patients in France). It is a late-onset form often presenting paroxysmal episodes of ataxia and/or diplopia. The disease progresses slowly, with an average increase of 0.10 points/year on the Friedreich's Ataxia Rating Scale (FARS) - Functional Staging and by 0.23 points/year on the Scale for the Assessment and Rating of Ataxia (SARA). To date, no treatment has been proven to be effective in these patients. Three open-label studies using 4-aminopyridine, have shown improvements in visual symptoms and gait in a total of 36 out of 44 patients, although these improvements were evaluated through diverse methodologies. In a subgroup of patients (n=7), administration of 4-aminopyridine resulted in a reduction in FARS - Functional Staging, ranging from 0.5 to 2 points. Notably, this beneficial effect rapidly disappearing in all patients stopping the drug. 4-aminopyridine, a potassium channel blocker, may involve restoration of cerebellar Purkinje cell rhythmic firing property, impaired with the loss of FGF14 function. Although these results appear very promising, the positive effect of 4-aminopyridine is reported only in restricted sample sizes and open-label experiences. Therefore, a robust clinical trial is necessary to provide the level of evidence required for a definitive conclusion on the benefit-risk of fampridine and before introducing the treatment into the regular patient clinical management.

Hence, to confirm the beneficial effect of 4-aminopyridine treatment, this study will compare fampridine 10 mg bid (sustained-release form) to placebo during a 3-month treatment in a randomized, double-blind, multicenter, placebo-controlled study, on functional handicap in SCA27B cerebellar ataxia patients.

ELIGIBILITY:
Inclusion Criteria:

* Genetic diagnosis of spinocerebellar ataxia SCA27B caused by an expansion ≥ 250 GAA repeats in the FGF14 gene
* At least 18 years of age
* SARA total score > 3 and score ≥ 1 on the "gait" item of the SARA scale.
* Physically able and expected to complete the trial as designed and having the ability to take oral medication
* Signature of informed consent
* Covered by social security

Exclusion Criteria:

* Hypersensitivity to fampridine
* Hypersensitivity to any excipients present in fampridine
* Serious systemic illnesses or conditions known for enhancing the side-effects of fampridine (i.e., creatinine clearance < 50 ml/min, hepatic insufficiency, medically significant heart conduction disorders such as occurrence of torsades de pointes or another severe ventricular arrhythmia, high-degree atrioventricular block (Mobitz II or complete), Brugada pattern, QTcF time of >480 msec in 3 consecutive ECG recordings taken at least 5 minutes apart, uncompensated cardiovascular disorder, epilepsy)
* Unstable, clinically significant neurologic (other than the disease being studied; eg, recurrent strokes), psychiatric, cardiovascular (eg, pulmonary arterial hypertension, cardiac valvulopathy, orthostatic hypotension/tachycardia), pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, immunologic, hematopoietic, or endocrine disease or other abnormality which may impact the ability of the participant to participate or potentially confound the study results.
* Patients with known recurrent, active, or chronic infections.
* Patients with prior history of seizure.
* Concurrent treatment with other medicinal products containing fampridine (4-aminopyridine).
* Concomitant use of Fampyra with medicinal products that are inhibitors or substrates of Organic Cation Transporter 2 (OCT2) for example, cimetidine.
* Participation in another clinical trial with an investigational drug or receipt of an investigational product within 12 weeks or 5 times the half-life of the product (whichever is longer) prior to Baseline visit
* Previous treatment with fampridine
* Patients considered at risk of suicidal behavior based on the Columbia-Suicide Severity Rating Scale (C-SSRS), defined as reporting suicidal ideation with intent to act (C-SSRS items 4 or 5) within the 6 months prior to randomization, or any suicidal behavior (including actual, aborted, or interrupted attempts) within the past 12 months.
* Pregnancy and breastfeeding (women in childbearing potential will have a urine pregnancy test at each visit)
* Sexual non abstinence or absence of effective contraception (for child-bearing aged women, contraception using highly effective methods (see section 6.2 of the protocol) for the duration of treatment and up to 7 days after the last dose of treatment)
* Inability to understand information about the protocol
* Legally incapacitated adults (e.g., individuals under legal protection such as guardianship or curatorship)
* Persons deprived of their liberty by judicial decision
* Other ataxic syndromes than SCA27B

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-10-21 (Actual); Primary Completion 2027-05-21 (Estimated); Study Completion 2027-05-21 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients showing an improvement of at least 0.5 point on the Friedreich's Ataxia Rating Scale (FARS) -Functional Staging at week 12 | At week 12

SECONDARY OUTCOMES:
Improvement of at least 0.5 point on the Friedreich's Ataxia Rating Scale (FARS) -Functional Staging at week 2 | At week 2
Variation in cerebellar syndrome assessed by the Scale for the assessment and rating of ataxia (SARA) at week 2 and week 12 | At week 2 and week 12
Variation in cerebellar syndrome assessed by the modified Friedreich Ataxia Rating Scale (mFARS) at week 2 and week 12 | At week 2 and week 12
Variation in cerebellar syndrome assessed by the Composite Cerebellar Functional Severity Score (CCFS score) at week 2 and week 12 | At week 2 and week 12
Variation in extracerebellar signs assessed by the Inventory of Non-Ataxia Signs (INAS) at week 12 | At week 12
Variation on Timed 25-foot walk (T25FW) at week 2 and week 12 | At week 2 and week 12
Variation in oculomotor signs assessed by the Scale for Ocular motor Disorders in Ataxia (SODA) at week 2 and week 12 | At week 2 and week 12
Variation in oculomotor signs assessed by oculomotor recording (OMR) at week 2 and week 12 | At week 2 and week 12
Variation in daily frequency of diplopia assessed on a Numerical Diplopia Rating Scale (NDRS) at week 2 and week 12 | At week 2 and week 12
Variation in daily living activities evaluated by the FARS -Activities of Daily Living scale (FARS-ADL) at week 12 | At week 12
Quality of life evaluated by the Patient Reported Outcome Measure of Ataxia (PROM-ATAXIA) questionnaire at week 12 | At week 12
Quality of life evaluated by the 36-Item Short Form Health Survey (SF-36) questionnaire at week 12 | At week 12
Patient's impression evaluated by the Patient Global Impression of change (PGI-C) at week 2 and week 12 | At week 2 and week 12
Clinician's impression evaluated by the Clinician Global Impression of Change (CGI-C) at week 2 and week 12 | At week 2 and week 12
Tolerance to the investigational drug | At week 2 and week 12
  Tolerance will be evaluated through clinical examination, blood analysis, and electrocardiogram (ECG) performed at Week 2 and Week 12. In addition, adverse events will be systematically recorded throughout the study period.
Clinical assessments at week 16, i.e. 4 weeks after treatment interruption | At week 16
Variation in cerebellar syndrome assessed by the FARS-Functional Staging at week 16, i.e. 4 weeks after treatment interruption | At week 16
Variation in cerebellar syndrome assessed by the SARA scale at week 16, i.e. 4 weeks after treatment interruption | At week 16
Variation in cerebellar syndrome assessed by the mFARS scale at week 16, i.e. 4 weeks after treatment interruption | At week 16
Variation in cerebellar syndrome assessed by the CCFS score at week 16, i.e. 4 weeks after treatment interruption | At week 16
Variation in extracerebellar signs assessed by the Inventory of Non-Ataxia Signs (INAS) at week 16, i.e. 4 weeks after treatment interruption | At week 16
Variation on Timed 25-foot walk (T25FW) at week 16, i.e. 4 weeks after treatment interruption | At week 16
Variation in oculomotor signs assessed by the Scale for Ocular motor Disorders in Ataxia (SODA) at week 16, i.e. 4 weeks after treatment interruption | At week 16
Variation in oculomotor signs assessed by oculomotor recording (OMR) at week 16, i.e. 4 weeks after treatment interruption | At week 16
Variation in daily frequency of diplopia assessed on a Numerical Diplopia Rating Scale (NDRS) at week 16, i.e. 4 weeks after treatment interruption | At week 16
Variation in daily living activities evaluated by the FARS -Activities of Daily Living scale at week 16, i.e. 4 weeks after treatment interruption | At week 16
Quality of life evaluated by the PROM-ATAXIA questionnaire at week 16, i.e. 4 weeks after treatment interruption | At week 16
Quality of life evaluated by the 36-Item Short Form Health Survey (SF-36) questionnaire at week 16, i.e. 4 weeks after treatment interruption | At week 16
Patient's impression evaluated by the Patient Global Impression of change (PGI-C) at week 16, i.e. 4 weeks after treatment interruption | At week 16
Clinician's impression evaluated by the Clinician Global Impression of Change (CGI-C) at week 16, i.e. 4 weeks after treatment interruption | At week 16

CONTACTS AND LOCATIONS:
Overall Officials: Giulia COARELLI, Principal Investigator — Assistance Publique - Hôpitaux de Paris (AP-HP)
Locations (9):
- France (9):
  - Neurology Department, CHU d'Angers, Angers
  - Genetics Department, CHU de Bordeaux, Bordeaux
  - Neurology and Gentics Department, CHU de Dijon, Dijon
  - Neurology Department, Hôpital Pierre Wertheimer Hospital, Lyon
  - Neurology Department, Gui De Chauliac Hospital, Montpellier
  - Genetics Department, Pitié-Salpêtrière University Hospital, Paris
  - Genetics Department, CHU de Rouen, Rouen
  - Neurology Department, CHRU de Strasbourg, Strasbourg
  - Neurology Department, CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.